CLINICAL TRIAL: NCT05691868
Title: An Open Label, Multi-Center, Single Arm Prospective Evaluation of Exactech Vantage Total Ankle System (Outside US)
Brief Title: Vantage Mobile Bearing Total Ankle System Post Market Clinical Follow-up (Outside US)
Status: Recruiting | Type: Observational
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: CR16-004
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis; Arthritis of Ankle; Failure, Prosthesis
MeSH Terms: conditions — Arthritis, Rheumatoid; Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of this study are to evaluate the performance and safety of the Vantage Mobile-Bearing Total Angle System. This study will follow subjects for a period of up to 10 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for total ankle arthroplasty
* Patient is at least 21 years of age
* Patient is likely to be available for follow-up out to 10 years
* Patient is willing to participate by complying with pre- and postoperative visit requirements
* Patient is willing and able to read and sign a study informed consent form

Exclusion Criteria:

* Patient with excessive bone loss at the ankle joint site
* Patient with severe osteoporosis
* Patient with complete talar avascular necrosis
* Patient with active osteomyelitis
* Patient with infection at the ankle site or infection at distant sites that could migrate to the ankle
* Patient with sepsis
* Patient with vascular deficiency in the involved limb
* Pateint with neuropathic joints
* Patient with neurological or musculoskeletal disease or loss of function that may adversely affect movement of the lower limb, gait, or weight bearing
* Patient with poor soft tissue coverage around the ankle
* Patient with Charcot arthropathy
* Previsous ankle arthrodesis with excision of the malleoli
* Excessive loads as cuased by activity or patient weight - per investigator discretion
* Skeletally immature patients (patient is less than 21 years if age at time of surgery)
* Patient with dementia
* Patient with known metal allergies
* Patients who are unwilling to provide informed consent
* Patients who are unlikely to be available for follow-up out to 10 years
* Patients who are not deemed suitable candidates for the subject device
* Patient is pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet eligibility criteria - Patients who consent to participate to return for follow-up visits out to 10 years or longer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
AOFAS | Through study completion, an average of 1 per year
  American Orthopedic Foot and Ankle Society Score (AOFAS) - Questionaire on pain (40 points), function (45 points) , and alignment (15 points) - 100 points score where 100 indicates a healthy midfoot
SMFA | Through study completion, an average of 1 per year
  Short Musculoskeletal Function Assessment (SMFA) Score - 46 items Patient questionnaire divided into two sections: 34 questions on patients function assessment and 12 questions covering how bothered patients are by their symptoms where 1 indicates no problems/no difficulty/ not bothered and 5 indicates unable to do/symptoms all the time/being greatly bothered
SF-36 | Through study completion, an average of 1 per year
  Short Form Health Survey (SF-36) Score - 36-item patient-reproted survey of patient health - It consists on 8 scales: Physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Each scale is transformed into a 0-100 scale where the lower score indicates the more disability and the higher score the lest disability
Sports Frequency Score | Through study completion, an average of 1 per year
  Sports Frequency Score - Level of sport activity in leisure time where 0 indicates "no sports activity" and 4 indicates "professional level of sports activity, elite athlete
VAS Pain score and Patient Satisfaction | Through study completion, an average of 1 per year
  Visual Analog Scale (VAS) Score - Range of scores from 0-100 to indicate level of pain - Higher score indicates greater pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Victor Valderrabano, MD, PhD, Principal Investigator — SWISS ORTHO CENTER Pain Clinic Basel; Mario Herrera- Perez, MD, PhD, Principal Investigator — Hospital Universitario de Canarias
Locations (2):
- Hospital Universitario de Canarias, Santa Cruz de Tenerife, Spain
- SWISS ORTHO CENTER Pain Clinic Basel, Basel, Switzerland